CLINICAL TRIAL: NCT01202838
Title: Bioactive Glass Composite Implants in Cranial Bone Reconstruction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Matti Peltola, adjunct professor, Turku University Hospital
Other Study IDs: MP125/2008
Record Dates: First submitted 2010-07-26; First posted 2010-09-16 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-09

CONDITIONS: Bone Substitutes
Keywords: Cranial bone reconstruction, composite

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Composite Implant: Subject receiving composite implant
  Interventions: Device: Composite Implant

INTERVENTIONS:
Device: Composite Implant — Subjects receiving composite implants

SUMMARY:
The purpose of this study is to study composites of bioactive glass and methylmetacrylate with glass fibre reinforcement in cranial bone defect reconstruction.

DETAILED DESCRIPTION:
Traditional skull and facial bone reconstructions with hard tissues have a long history with good clinical outcomes. However, they have certain disadvantages. The benefits of synthetic materials are the avoidance of donor-site morbidity and scars, but also shorter hospitalization time, lower expenses and known composition. Custom-made skull bone implant can produced based on patients clinical need utilizing rapid prototyping technologies. This will result in very high accuracy of the form of the skull defect.

Polymethylmetacrylate (PMMA) is one of the most widely used alloplastic material in surgery. Bioactive glass S53P4 (BAG) particles have been used in various clinical indications. BAG was added to composite implant of PMMA with glass fibre reinforcement to enhance bone ingrowth to implant, and to utilize BAG's antimicrobial effects. Ten patients cranial defects are treated with composite implants.

ELIGIBILITY:
Inclusion Criteria:

* patients with cranial bone defect larger than 4x4 cm after trauma or tumor surgery
* patient signs written study consent

Exclusion Criteria:

* patient is unlikely to adhere to study procedures
* patient has a disease or condition that in the opinion of investigator is contraindicating participation
* patient is participating another medical device or drug trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of Turku university hospital needing cranial bone defect reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2008-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Clinical success | 3 years
  Clinical success is evaluated using clinical and radiographic examination, and blood count.

CONTACTS AND LOCATIONS:
Overall Officials: Matti J Peltola, MD, PhD, DDS, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

REFERENCES:
- [Background] Peltola MJ, Aitasalo KM, Aho AJ, Tirri T, Suonpaa JT. Long-term microscopic and tissue analytical findings for 2 frontal sinus obliteration materials. J Oral Maxillofac Surg. 2008 Aug;66(8):1699-707. doi: 10.1016/j.joms.2007.11.020. No abstract available. PMID 18634960
- [Background] Peltola M, Aitasalo K, Suonpaa J, Varpula M, Yli-Urpo A. Bioactive glass S53P4 in frontal sinus obliteration: a long-term clinical experience. Head Neck. 2006 Sep;28(9):834-41. doi: 10.1002/hed.20436. PMID 16823870
- [Background] Tuusa SM, Peltola MJ, Tirri T, Puska MA, Roytta M, Aho H, Sandholm J, Lassila LV, Vallittu PK. Reconstruction of critical size calvarial bone defects in rabbits with glass-fiber-reinforced composite with bioactive glass granule coating. J Biomed Mater Res B Appl Biomater. 2008 Feb;84(2):510-9. doi: 10.1002/jbm.b.30898. PMID 17618510
- [Background] Lepparanta O, Vaahtio M, Peltola T, Zhang D, Hupa L, Hupa M, Ylanen H, Salonen JI, Viljanen MK, Eerola E. Antibacterial effect of bioactive glasses on clinically important anaerobic bacteria in vitro. J Mater Sci Mater Med. 2008 Feb;19(2):547-51. doi: 10.1007/s10856-007-3018-5. Epub 2007 Jul 10. PMID 17619981
- [Background] Munukka E, Lepparanta O, Korkeamaki M, Vaahtio M, Peltola T, Zhang D, Hupa L, Ylanen H, Salonen JI, Viljanen MK, Eerola E. Bactericidal effects of bioactive glasses on clinically important aerobic bacteria. J Mater Sci Mater Med. 2008 Jan;19(1):27-32. doi: 10.1007/s10856-007-3143-1. Epub 2007 Jun 14. PMID 17569007